CLINICAL TRIAL: NCT02578498
Title: Glucagon Efficiency After High and Low Carbohydrate Diet
Acronym: HiLoCarb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Danish Diabetes Academy (Other)
Responsible Party: Principal Investigator, Ajenthen Ranjan, MD, PhD student, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: H-15009662
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2015-10

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: glucagon; Carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High carbohydrate diet (Placebo Comparator): high carbohydrate intake
  Interventions: Dietary Supplement: Low carbohydrate intake
- Low carbohydrate diet (Active Comparator): low carbohydrate intake
  Interventions: Dietary Supplement: High carbohydrate intake

INTERVENTIONS:
Dietary Supplement: High carbohydrate intake — Carbohydrate intake < 50 gram
  Arms: Low carbohydrate diet
Dietary Supplement: Low carbohydrate intake — Carbohydrate intake > 250 gram
  Arms: High carbohydrate diet

SUMMARY:
No studies have investigated if the dietary composition of carbohydrate influences the glycaemic effect of single and multiple boluses of subcutaneous low-dose glucagon. Further, the recommended diet composition to patients with type 1 diabetes has not been thoroughly validated. Many patients with type 1 diabetes practice low carbohydrate eating patterns due to the assumption that this diet can reduce fluctuations in plasma glucose. Before glucagon can be used as an add-on to intensive insulin treatment, these aspects need to be elucidated. The purpose of this study is to determine, whether diet composition of carbohydrate affects the glycogen stores in the liver and affects the glucose response of glucagon during hypoglycaemia.

HYPOTHESIS: In patients with type 1 diabetes, the glucose response of a single bolus of low-dose glucagon is not associated with diet carbohydrate content.

AIM: The aim is to investigate how one week of high- compared to low-carbohydrate diet influence the glycaemic response of low-dose glucagon in patients with insulin pump treated type 1 diabetes. The secondary aim is to investigate how two dietary intervention weeks differ in the incidence of hypoglycaemia, postprandial hyperglycaemia, and daily glucose excursions.

DESIGN:A non-blinded two-way cross-over, randomized study will be conducted. After participants have given an informed consent, they will go through four steps: 1) screening visit 2) Run-in period, 3) first meal intervention for one week finalizing with one study visit and 4) second meal intervention for one week finalizing with another study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* T1D ≥ 3 year
* BMI 20-27 kg/m2
* CSII ≥ 1 year
* HbA1c < 69 mmol/mol (8.5 %)
* C-peptide negative (< 60 pmol/l)
* Hypoglycemia awareness (self-reported)
* Use of carbohydrate counting and the insulin pump bolus calculator for all meals

Exclusion Criteria:

* Allergy or intolerance to lactose or Glucagen®(Novo Nordisk, Bagsværd, DK)
* Impaired renal function (eGFR < 60 ml/min/1.73m2)
* Liver disease with ALAT > 2.5 times the upper limit of the reference interval
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods.
* Inability to understand the patient information and to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incremental area under the glucose curve | 0-240 minutes
Peak glucose value | within 240 minutes

SECONDARY OUTCOMES:
Glucagon concentration | 0-240 min.
  Blood samples
Insulin concentration | 0-240 min.
  Blood samples
Triglycerides concentration | 0-240 min.
  Blood samples
Katekolamine concentration | 0-240 min.
  Blood samples
Ketone bodies concentration | 0-240 min.
  Blood samples
Free fatty acids concentration | 0-240 min.
Nausea | 0-240 min.
  Visual analog scale
Headache | 0-240 min.
  Visual analog scale
Hypoglycemia symptoms | 0-240 min.
  Visual analog scale
Vomit | 0-240 min.
  Occurence
Plasma glucose variation | Two weeks
  A continuous glucose monitor register daily glucose variation levels for two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, MD, DMSc, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Ranjan A, Schmidt S, Damm-Frydenberg C, Steineck I, Clausen TR, Holst JJ, Madsbad S, Norgaard K. Low-Carbohydrate Diet Impairs the Effect of Glucagon in the Treatment of Insulin-Induced Mild Hypoglycemia: A Randomized Crossover Study. Diabetes Care. 2017 Jan;40(1):132-135. doi: 10.2337/dc16-1472. Epub 2016 Oct 21. PMID 27797928